CLINICAL TRIAL: NCT05509140
Title: Clinical Analysis of 12 Cases of Juvenile Dermatomyositis Treated With Methylprednisolone Repeated Intermittent Pulse Combined With Mycophenolate Mofetil
Brief Title: Clinical Analysis of Juvenile Dermatomyositis Patients
Status: Completed | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, SiRui Yang, professor, The First Hospital of Jilin University
Other Study IDs: 2020-613
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Juvenile Dermatomyositis
Keywords: intravenous methylprednisolone repeated intermittent pulse; mycophenolate mofetil
MeSH Terms: conditions — Dermatomyositis | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation — investigate the clinical effectivity of intravenous methylprednisolone repeated intermittent pulse combined with mycophenolate mofetil in the treatment of newly diagnosed juvenile dermatomyositis

SUMMARY:
This study aimed to investigate the clinical effectivity of intravenous methylprednisolone repeated intermittent pulse combined with mycophenolate mofetil in the treatment of newly diagnosed juvenile dermatomyositis.

DETAILED DESCRIPTION:
Reviewed the clinical data of 12 juvenile dermatomyositis patients, from January 2014 to January 2017, hospitalized and treated with intravenous methylprednisolone repeated intermittent pulse combined with mycophenolate mofetil

ELIGIBILITY:
Inclusion Criteria:

1. patients with age of JDM onset <16 years
2. newly treated cases
3. no contraindications to corticosteroids
4. provide signed informed consent form
5. regular follow-up for more than 30 months.

Exclusion Criteria:

1. patients with serious complications of heart, liver and kidney
2. patients with a history of contraindications and/or allergies to GC
3. patients who underwent treatment before admission
4. patients who failed to regularly follow-up
5. patients with positive anti-melanoma differentiation-associated gene 5 (MDA5) antibodies

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients who meet the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in CMAS score | 1, 3, 6, 12, 18, 24 and 36 months
  CMAS score is an index to assess the disease activity of JDM

SECONDARY OUTCOMES:
Changes from baseline of the patient's height percentile in the same age and sex crowd. | 1, 3, 6, 12, 18, 24 and 36months
  the patient's height percentile in the same age and sex crowd is one of safety evaluation indicators.
Changes from baseline of the patient's weight percentile in the same age and sex crowd. | 1, 3, 6, 12, 18, 24 and 36months
  the patient's weight percentile in the same age and sex crowd is one of safety evaluation indicators.
intraocular pressure | 1, 3, 6, 12, 18, 24 and 36months
  the patient's intraocular pressure is one of safety evaluation indicators.
triglycerides | 1, 3, 6, 12, 18, 24 and 36months
  the patient's triglycerides is one of safety evaluation indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Sirui Yang, doctor, Principal Investigator — The First Hospital of Jilin University